CLINICAL TRIAL: NCT06256120
Title: Effects of Peroperative Liberal and Restrictive Fluid Regimens on Protection From Postoperative Acute Kidney Injury in Patients Undergoing Partial or Radical Nephrectomy; Randomized Controlled Trial
Brief Title: Effect of Fluid Regimen on Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Eylem Yaşar, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Mugla SKU
Record Dates: First submitted 2023-12-26; First posted 2024-02-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Nephrectomy; Acute Kidney Injury; Fluid Therapy
Keywords: Nephrectomy; Acute Kidney Injury; Cystatin; Fluid treatment
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into two groups: restrictive and liberal fluid replacement groups. 3 ml/kg/hour Ringer's lactate (RL) solution will be given to the group that will receive restrictive fluid replacement (Group R), and 7 ml/kg/hour RL solution will be given to the group that will receive liberal fluid regimen (Group L). Patients in both groups will receive 1.5 ml/kg/hour crystalloid fluid replacement on postoperative day 1, and oral intake will be increased on day 2.
  Serum creatinine, GFR and blood urea nitrogen (BUN) values will be measured in all patients before surgery and 48 hours after removal of the renal pedicle clamp. Patients' blood and blood product replacement, vasopressor and inotrope needs will be recorded. Serum cystatin C level will be measured by taking serum samples before the surgery and at the 48th hour postoperatively.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and those evaluating blood samples will not know which group they are in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R- fluid group (Experimental): The group to which restrictive fluid replacement will be applied (Group R); 3 ml/kg/hour Ringer lactate (RL) solution will be given.
  Interventions: Diagnostic Test: Restrictive
- L- fluid group (Experimental): 7 ml/kg/hour RL solution will be given to the group that will receive a liberal liquid regimen (Group L).
  Interventions: Diagnostic Test: Liberal

INTERVENTIONS:
Diagnostic Test: Restrictive — 3 mL/kg/hour Ringer Lactate will be given peroperatively to the restrictive group (Group R).
  Arms: R- fluid group
Diagnostic Test: Liberal — 7 ml/kg/hour Ringer Lactate will be given peroperatively to the liberal group (Group L).
  Arms: L- fluid group

SUMMARY:
Postoperative acute kidney injury (AKI) is an important surgical complication that increases hospital stay and mortality when it occurs after kidney surgery. Studies investigating the effects of restrictive or liberal fluid regimen on postoperative AKI during radical/partial nephrectomy have given controversial results. It is important to recognize AKI early so that supportive treatments can be started early. Serum creatinine level, which is frequently used in the detection of AKI, increases late and causes a delay in diagnosis. It has been reported that cystatin C level increases earlier than creatinine in the diagnosis of AKI, so it can be used for early diagnosis.

DETAILED DESCRIPTION:
Hypovolemia and organ dysfunction may occur as a result of giving too little fluid during the operation; Giving too much fluid can also cause edema and organ damage. AKI, which develops after kidney surgery, is an important surgical complication and its incidence varies between 5.5% and 34%. Kidney damage is initially subclinical, and its detection is delayed with current diagnostic tools. Due to increased microvascular permeability as a result of excessive fluid administration during the operation, edema in organ tissues and systems may increase infection rates and kidney damage. In a study in which restrictive and free fluid was applied during abdominal aortic aneurysm surgery, they showed that there was deterioration in renal endothelial function in the liberal group; They found that the urine albumin/creatinine ratio increased. In another study, they reported that serum creatinine levels decreased on the first day in patients who underwent colorectal surgery in the group where they applied a liberal fluid regimen; However, they reported that they could not find a significant difference between them and the restrictive group on the following days. It has been shown that restrictive and liberal fluid management applied during abdominal surgery have no effect on renal functions. Although there are few studies in the literature showing that restrictive and liberal fluid regimens applied during abdominal operations affect postoperative renal functions; There are no studies investigating the ideal intraoperative fluid replacement in nephrectomy patients.

It is known that the serum creatinine level, which is routinely used to monitor renal functions, increases late and has poor sensitivity. The reason for this is that it begins to increase 48-72 hours after kidney damage begins and when 50% of functional neurons are lost. Cystatin C, produced by all nucleated cells, is freely filtered by the glomerulus and reabsorbed in the proximal tubule. It is not secreted by renal tubules and does not vary depending on gender, race, weight, changes in muscle mass and nutrition. Serum cystatin C is a biomarker that reflects glomerular filtration rate (GFR) well and can diagnose AKI more accurately than creatinine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II-III,
* The opposite kidney is in normal function

Exclusion Criteria:

* Those who are planned for bilateral partial nephrectomy,
* Patients with preoperative chronic kidney disease,
* Those using preoperative medications known to cause renal toxicity such as aminoglycosides, aspirin and angiotensin converting enzyme inhibitors,
* Coronary artery disease
* Congestive heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
rate of acute renal failure | 48 hour
  To determine whether the restrictive or liberal fluid regimen applied during partial or radical nephrectomy surgery causes acute renal failure in the early postoperative period.

SECONDARY OUTCOMES:
Creatinine | 48 hour
  Comparison of creatinine elevation between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Yasar, M.D, Principal Investigator — Mugla Sitki Kocman Training and Research Hospital
Locations (1):
- Mugla Sitki Kocman Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data, except patient names, will be shared with the editor upon request after the article is accepted.

REFERENCES:
- [Derived] Yasar E, Toker MK, Saruhan E, Gursoy C. Impact of liberal versus restrictive fluid management on acute kidney injury after nephrectomy: a randomised controlled trial with cystatin C evaluation. BMC Urol. 2025 Oct 27;25(1):270. doi: 10.1186/s12894-025-01954-w. PMID 41146149